CLINICAL TRIAL: NCT00878475
Title: Quantitative Capnometry and Nt-proBNP in Differentiating of Acute Dyspnea in Pre-Hospital Emergency Setting
Brief Title: Dyspnea and Biomarkers in a Prehospital Setting
Status: Completed | Type: Observational
Sponsor: Community Healthcare Center dr. Adolf Drolc Maribor (HCM) (Other)
Responsible Party: Prof.Štefek Grmec, MD, PhD, Health Center Maribor, Emergency Medicine center
Other Study IDs: grmec62
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Dyspnea; Heart Failure; Asthma; COPD
Keywords: Quantitative Capnometry; N-Terminal Pro-Brain Natriuretic Peptide; Acute Heart Failure; Diagnostic Accuracy
MeSH Terms: conditions — Dyspnea; Heart Failure; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group with obstructive causes of dyspnea: Criteria for clinical assessment of severe asthma (diffuse polyphonic bilateral and particular expiratory wheezes, chest tightness, shortness of breath, using accessory muscles of breathing, signs of hyperinflation, atopic condition, personal or family history of asthma, tachypnea, previous asthma and asthma medications, and the value of modified Boston criteria for HF ≤ 5) and criteria for chronic obstructive pulmonary disease (COPD) exacerbation (history of COPD, COPD medications, cough, worsening dyspnea, increased sputum production and volume, increased sputum purulence, rhonchi and rales, modified Boston criteria for HF ≤ 5)
- Heart failure group: The investigators protocol for clinical assessment of HF-related acute dyspnea (the prehospital clinical assessment for HF) was designed based on Boston (13) and Framingham criteria for HF (14) (Table 1). The investigators did not use certain criteria from the original protocols, which were not available in the prehospital setting (e.g., chest radiography).

SUMMARY:
In patients presenting with acute dyspnea in a pre-hospital setting, the early and correct diagnosis may present a significant clinical challenge. Physical examination, chest radiography, electrocardiography, and standard biological tests often fail to accurately differentiate heart failure (HF) from pulmonary causes of dyspnea. Timely differentiation of HF from other causes of dyspnea may permit the early institution of appropriate medical therapy. Brain natriuretic peptide (BNP) and amino-terminal pro-brain natriuretic peptide (NT-proBNP) have been proposed as early markers of HF and demonstrated to be useful for diagnosing and excluding HF in the emergency department. A combination of BNP or NT-proBNP testing and standard clinical assessment has been suggested to be superior to either tool used in isolation. Some previous studies have also suggested that quantitative capnometry (QC) may be useful in differentiating between cardiac and obstructive causes of respiratory distress. Therefore, the investigators hypothesized that a new combination of NT-proBNP testing, standard clinical assessment, and partial pressure of end-tidal CO2 (PetCO2) would optimize evaluation and differentiation of acute dyspnea in a pre-hospital setting.

The aim of this study was to determine the accuracy of combination of QC, NT-proBNP, and clinical assessment in differentiating acute HF from obstructive pulmonary disease (COPD/asthma) as a cause of acute dyspnea in pre-hospital emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* patient had to present with shortness of breath as the primary complaint (defined as either the sudden onset of dyspnea without history of chronic dyspnea or an increase in the severity of chronic dyspnea)

Exclusion Criteria:

* age <18 years
* history of renal insufficiency, trauma, severe coronary ischemia (unless patient's predominant presentation was dyspnea), and other causes of dyspnea:

  * pneumonia
  * pulmonary embolism
  * carcinoma
  * pneumothorax
  * pleural effusion
  * intoxications (drugs)
  * anaphylactic reactions
  * upper airway obstruction
  * bronchial stenosis
  * gastroesophageal reflux disorder
* according to the history, clinical status, and additional laboratory tests available in pre-hospital setting (D-dimer, troponin, C-reactive protein)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: During the period of the study, 546 consecutive patients with acute dyspnea were treated by emergency teams (emergency physician, register nurse, and medical technician/driver in an ambulance-car or at pre-hospital emergency medical center). After pre-hospital care, all patients were admitted to the University Clinical Center Maribor and followed until discharge.
  To be eligible for the study, a patient had to present with shortness of breath as the primary complaint (defined as either the sudden onset of dyspnea without history of chronic dyspnea or an increase in the severity of chronic dyspnea).
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Štefek Grmec, Prof,MD,PhD, Principal Investigator — Health Center, Center for emergency Medicine Maribor
Locations (1):
- Health Center Maribor, Center for Emergency Medicine, Maribor, Slovenia

REFERENCES:
- [Derived] Klemen P, Golub M, Grmec S. Combination of quantitative capnometry, N-terminal pro-brain natriuretic peptide, and clinical assessment in differentiating acute heart failure from pulmonary disease as cause of acute dyspnea in pre-hospital emergency setting: study of diagnostic accuracy. Croat Med J. 2009 Apr;50(2):133-42. doi: 10.3325/cmj.2009.50.133. PMID 19399946